CLINICAL TRIAL: NCT06112314
Title: A Phase 3 Randomized, Controlled Study of IMC-F106C Plus Nivolumab Versus Nivolumab Regimens in HLA-A*02:01-Positive Participants With Previously Untreated Advanced Melanoma (PRISM-MEL-301
Brief Title: IMC-F106C Regimen Versus Nivolumab Regimens in Previously Untreated Advanced Melanoma (PRISM-MEL-301)
Acronym: PRISM-MEL-301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMC-F106C-301; 2023-505306-42 (Other: EU CT Number)
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Brenetafusp Low Dose + Nivolumab (Experimental): Participants receive brenetafusp Low Dose once weekly (QW) for the first 13 weeks, then every 2 weeks (Q2W) through Week 51, and then every 4 weeks (Q4W). Nivolumab is given Q4W.
  Interventions: Drug: Brenetafusp; Drug: Nivolumab
- Arm B: Brenetafusp High Dose + Nivolumab (Experimental): Participants receive brenetafusp High Dose once weekly (QW) for the first 13 weeks, then every 2 weeks (Q2W) through Week 51, and then every 4 weeks (Q4W). Nivolumab is given Q4W.
  Interventions: Drug: Brenetafusp; Drug: Nivolumab
- Arm C: Nivolumab OR Nivolumab + Relatlimab (Active Comparator): Participants receive nivolumab 480 mg monotherapy, or nivolumab 480 mg + relatlimab 160 mg, Q4W.
  Interventions: Drug: Nivolumab; Drug: Nivolumab + Relatlimab

INTERVENTIONS:
Drug: Brenetafusp — Soluble PRAME-specific T cell receptor with anti-CD3 scFV concentrate for solution for intravenous (IV) infusion at a unit dose of 0.2 mg/mL.
  Other Names: IMC-F106C
  Arms: Arm A: Brenetafusp Low Dose + Nivolumab; Arm B: Brenetafusp High Dose + Nivolumab
Drug: Nivolumab — Concentrate for solution for infusion at a unit dose of 10 mg/mL.
  Other Names: OPDIVO
Drug: Nivolumab + Relatlimab — Concentrate for solution for infusion at a unit dose of 16 mg/mL.
  Other Names: OPDUALAG
  Arms: Arm C: Nivolumab OR Nivolumab + Relatlimab

SUMMARY:
This is a phase 3, randomized, controlled study of brenetafusp (IMC-F106C) plus nivolumab compared to standard nivolumab regimens in HLA-A*02:01-positive participants with previously untreated advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be HLA-A*02:01-positive
* Participants must have histologically confirmed Stage IV or unresectable Stage III melanoma
* Archived or fresh tumor tissue sample that must be confirmed as adequate
* Participants must have measurable disease per RECIST 1.1
* Participant must have BRAF V600 mutation status determined
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Male and female participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control from the study screening date until 5 months after the final dose of study intervention

Exclusion Criteria:

* Participants with a history of a malignant disease other than those being treated in this study
* Participants with untreated, active, or symptomatic central nervous system (CNS) metastases or carcinomatous meningitis
* Hypersensitivity to IMC-F106C, nivolumab, relatlimab, or any associated excipients
* Participants with clinically significant pulmonary disease or impaired lung function
* Participants with clinically significant cardiac disease or impaired cardiac function
* Participants with active autoimmune disease requiring immunosuppressive treatment
* Participants with any medical condition that is poorly controlled or that would, in the Investigator's or Sponsor's judgment, adversely impact the participant's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results
* Participants who received prior systemic anticancer therapy for unresectable or metastatic melanoma
* Participants with a history of a life-threatening AE related to prior anti-PD-(L)1 or anti-LAG-3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-10-16 (Estimated); Study Completion 2027-10-16 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to ~45 months
  PFS as assessed by blinded independent central review (BICR) according to Response Evaluation Criteria in Solid Tumours (RECIST 1.1).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~57 months
  OS is the time from randomization to time of death from any cause.
Overall Response Rate (ORR) | Up to ~45 months
  ORR as assessed by BICR according to RECIST 1.1.
Number of Participants Experiencing ≥1 Adverse Event (AE) | Up to ~57 months
  An AE is defined as the appearance of (or worsening of any pre-existing) undesirable sign, symptom, or medical condition that occur in the study.
Number of Participants Experiencing ≥1 Serious Adverse Event (SAE) | Up to ~57 months
  An SAE is any untoward medical consequence that results in death; requires inpatient hospitalization or prolongs existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or any other important medical event in the opinion of the Investigator.
Number of Participants Experiencing a Dose Interruption, Reduction, or Discontinuation | Up to ~45 months
  The number of participants with a dose interruption, reduction, or discontinuation due to AE will be reported.
Maximum Plasma Concentration (Cmax) of IMC-F106C | Day 1 of Weeks 1, 2, and 3: Predose and 0.5 and 4 hours postdose
  The Cmax of IMC-F106C will be reported.
Incidence of anti-IMC-F106C Antibodies | Up to ~45 months
  The incidence of anti-IMC-F106C antibodies, including neutralizing antibodies, will be reported.
Association between PFS and Intra-Tumor Immune Cells | Up to ~45 months
  The potential association between the effect of IMC-F106C on efficacy and intra-tumor environment will be explored. Intra-tumor environment is estimated as the ratio of CD3+ to CD163+ cells and the correlation with PFS will be estimated by the hazard ratio (+/- 95% CI) from a Cox model. This analysis will be restricted to subjects randomized to receive IMC-F106C.
Health-Related Quality of Life | Up to ~45 months
  The change from baseline over time and between treatments of health-related quality of life will be reported.

CONTACTS AND LOCATIONS:
Locations (173):
- United States (28):
  - University of Arizona, Tucson, Arizona
  - University of California - San Diego, La Jolla, California
  - The Angeles Clinic and Research Institute- West Los Angeles, Los Angeles, California
  - ESC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Stanford Cancer Institute - Stanford Cancer Center Palo Alto, Palo Alto, California
  - Saint John's Health Center - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - UConn Health-Farmington (University of Connecticut Health Center (UCHC)), Farmington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami Health System-Sylvester Comprehensive Cancer Center-Miami, Miami, Florida
  - Northwestern University - Robert H. Lurie Comprehensive Cancer Center - NMDTI, Chicago, Illinois
  - The University of Kansas Cancer Center (KUCC) - Westwood, Westwood, Kansas
  - St. Elizabeth Healthcare - Edgewood, Edgewood, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health Cancer Institute, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Spartanburg Regional Healthcare System - Spartanburg Medical Center (SMC), Spartanburg, South Carolina
  - Sarah Cannon Research Institute: USA/TN, Nashville, Tennessee
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - UVA Health-UVA Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Swedish Medical Center - Swedish Cancer Institute (SCI) - First Hill Campus, Seattle, Washington
- Argentina (5):
  - Sanatorio Finochietto, Caba, Buenos Aires
  - Clínica Adventista Belgrano - Sector Investigación, Caba, Buenos Aires
  - Instituto Alexander Fleming, CABA
  - CEMAIC (Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Clinica Viedma, Viedma
- Australia (8):
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Gallipoli Medical Research Foundation (Greenslopes Private Hospital), Greenslopes, Queensland
  - Linear Clinical Research, Nedlands, Western Australia
  - One Clinical Research - Nedlands, Nedlands, Western Australia
  - Austin Hospital, Heidelberg
  - Peter MacCallum Cancer Centre, North Melbourne
  - University of Sydney - Melanoma Institute Australia (MIA) - The Poche Centre, Wollstonecraft
  - The University of Queensland (UQ) - Princess Alexandra Hospital (PAH), Woolloongabba
- Austria (3):
  - LKH - Universitaetsklinikum Graz, Graz
  - Universitätsklinikum St. Pölten, Pölten
  - Paracelsus Medizinischen Privatuniversitaet - SALK - Universitaetsklinik fuer Dermatologie - EB-Haus Austria, Salzburg
- Belgium (5):
  - Universite Libre de Bruxelles (ULB)-Institut Jules Bordet, Anderlecht
  - AZ Sint-Jan Brugge-Oostende AV-Campus Sint-Jan, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc - Institut Roi Albert II, Brussels
  - UZ Leuven, Leuven
- Brazil (14):
  - Centro de Pesquisa Clinica em Oncologia - Oncosite, Ijuí, Rio Grande do Sul
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa Ltda, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos - Hospital de Amor, Barretos
  - Hospital Sirio-Libanes (HSL) - Centro de Oncologia - Brasilia, Brasília
  - Centro de Pesquisas Oncologicas (CEPON), Florianópolis
  - Oncocentro Sao Carlos Hospital, Fortaleza
  - A.C.Camargo Cancer Center - Centro Internacional de Pesquisa (CIPE), Liberdade
  - Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre
  - Pontificia Universidade Catolica do Rio Grande do Sul (PUCRS) - Hospital Sao Lucas - Centro de Pesquisa Clinica (CPC), Porto Alegre
  - National Cancer Institute, Rio de Janeiro
  - Instituto Américas - Instituto de Educação Pesquisa e Gestão em Saúde Oncosite, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo (ICESP), São Paulo
  - Hospital 9 de Julho, São Paulo
  - Faculdade de Medicina de Sao Jose do Rio Preto-SP (FAMERP) - Hospital de Base (HB) - Centro Integrado de Pesquisa (CIP), São Paulo
- Bulgaria (4):
  - Uni Hospital, Panagyurishte
  - Complex Oncology Center - Plovdiv Ltd., Plovdiv
  - University Hospital Tsaritsa Yoanna (ISUL) (Queen Giovanna University Hospital), Sofia
  - Regina Life Clinic, Sofia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Cross Cancer Institute, Edmonton
- Czechia (3):
  - Fakultni Nemocnice Hradec Kralove (FNHK) - Klinika Onkologie a Radioterapie, Hradec Králové
  - Fakultni Nemocnice Olomouc (FNOL), Olomouc
  - Sanatorium Profesora Arenbergera, Prague
- Kobenhavns Universitet - Herlev Hospital (Amtssygehuset i Herlev), Herlev, Denmark
- France (13):
  - Hôpital de la Timone, Marseille, Cedex
  - Oncopole Claudius Regaud- Institut Universitaire du Cancer de Toulouse, Toulouse, Cedex
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopitaux Universitaires Paris Seine-Saint-Denis - Hopital Avicenne, Bobigny
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Ambroise-Pare, Boulogne-Billancourt
  - UNICANCER-Centre Francois Baclesse (CFB), Caen
  - CHU de Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Centre Hospitalier Universitaire de Lille (CHU Lille)-Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hotel-Dieu, Nantes
  - Hospital Saint Louis, Paris
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rouen (CHU de Rouen) - Hopital Charles-Nicolle, Rouen
  - Hopital Robert Debre, Valence
  - Institut Gustave Roussy (IGR) Service de Dermatolgie, Villejuif
- Germany (14):
  - Charite-Universitaetsmedizin Berlin - Campus Charite Mitte (CCM) - Klinik fuer Dermatologie Venerologie und Allergologie - Hauttumorcentrum Charite (HTCC), Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Helios Klinikum Erfurt - Klinik fuer Hautkrankheiten und Allergologie, Erfurt
  - Universitaetsklinikum Essen, Essen
  - Johann Wolfgang Goethe-Universitaet Frankfurt am Main - Klinik fuer Dermatologie, Venerologie und Allergologie, Frankfurt
  - Justus-Liebig-Universitaet Giessen - Klinik fuer Dermatologie und Andrologie, Giessen
  - University of Hamburg, Hamburg
  - Elbe Kliniken Stade - Hautkrebszentrum Buxtehude, Hamburg
  - Universitaetsklinikum Heidelberg (UKHD) - Hautklinik, Heidelberg
  - Universitaetsklinikum Leipzig - Klinik fuer Dermatologie, Venerologie und Allergologie, Leipzig
  - Johannes Wesling Klinikum Minden, Minden
  - LMU Klinikum - Klinik und Poliklinik fur Dermatologie und Allergologie, Munich
  - Universitaetsklinikum Tuebingen (UKT) - Zentrum fuer Dermatoonkologie - Hautklinik, Tübingen
  - Universitaetsklinikum Wuerzburg - Klinik und Poliklinik fuer Dermatologie Venerologie und Allergologie, Würzburg
- Hungary (3):
  - Semmelweis Egyetem Általános Orvostudományi Kar, Budapest
  - Pecsi Tudomanyegyetem (PTE) (University of Pecs), Pécs
  - Szegedi Tudomanyegyetem (University of Szeged), Szeged
- Italy (13):
  - Istituto Tumori Giovanni Paolo II - Ospedale Oncologico di Bari, Bari
  - Humanitas Gavazzeni (Cliniche Gavazzeni S.p.A), Bergamo
  - IRCCS Istituto Scientifico Romagnolo per lo Studio dei Tumori "Dino Amadori" Srl (IRST), Meldola
  - Istituto Europeo di Oncologia (IEO) (European Institute of Oncology), Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori - Milano, Milan
  - Istituto Nazionale Tumori (INT) "Fondazione G. Pascale" di Napoli, Napoli
  - Istituto Oncologico Veneto (IOV) IRCCS, Padua
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Sanitaria Locale di Biella (ASL BI) - Ospedale degli Infermi, Ponderano
  - National Cancer Institute Regina Elena, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - " Azienda Ospedaliera Universitaria Senese - Policlinico Santa Maria Alle Scotte - Clinica Immunoterapia Oncologica", Siena
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- Poland (4):
  - Centrum Onkologii im. Prof. Franciszka Łukaszczyka, Bydgoszcz
  - Klinika Onkologii i Radioterapii Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne Pratia Poznań - Skorzewo, Skorzewo
  - Klinika Nowotworów Tkanek Miękkich, Kości i Czerniaków, Warsaw
- Romania (3):
  - L'Institute Oncologique Prof. Dr. Ion Chiricuta (IOCN) (The Oncology Institute Prof. Dr. Ion. Chiricuta), Cluj-Napoca
  - Sf Nectarie Oncology Center, Craiova
  - Victoria Hospital (Centrul de oncologie Euroclinic SRL) (Centrul De Oncologie Medicala) (Euroclinic Onchology Center), Iași
- Spain (23):
  - Universidad de Cantabria (UC) - Hospital Universitario Marques de Valdecilla (HUMV), Santander, Cantabria
  - Universidad de Murcia - Hospital Universitario Virgen de la Arrixaca (HUVA), El Palmar, Murcia
  - Complejo Hospitalario Universitario A Coruna (CHUAC), A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Dexeus, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves (HUVN), Granada
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN) - Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Universidad Complutense de Madrid (UCM)-Hospital Universitario 12 de Octubre (H12O), Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN) - Pamplona, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto de Investigacion Sanitaria (INCLIVA) (Institute of Health Research Hospital Clinic of Valencia), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
  - Servicio Aragones de Salud - Hospital Universitario Miguel Servet (HUMS), Zaragoza
- Sweden (5):
  - Sahlgrenska Akademin - Institutionen for Kliniska Vetenskaper (Institute of Clinical Sciences), Gothenburg
  - Lanssjukhuset Ryhov - Onkologiska Kliniken, Jönköping
  - Skanes Universitetssjukhus - Lund - Onkologiska Klinik, Lund
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala Universitet - Akademiska Sjukhuset (Uppsala University Hospital), Uppsala
- UniversitaetsSpital Zuerich - Dermatologische Klinik, Zurich, Switzerland
- Turkey (Türkiye) (13):
  - Memorial Saglik Grubu - Memorial Ankara Hastanesi, Çankaya, Ankara
  - Medical Park Hastaneler Grubu - I.A.U. VM Medical Park Florya, Antalya, Campus
  - Medical Park Gaziantep Hastanesi, Şehitkamil, Gaziantep
  - Memorial Saglik Grubu - Memorial Bahcelievler Hastanesi, Bahçelievler, Istanbul
  - Ege Universitesi Tip Fakultesi (Ege University Faculty of Medicine), Bornova, İzmir
  - Izmir Ekonomi Universitesi Medikal Point Hastanesi, Cordaleo, İzmir
  - Kanser Enstitusu (Hacettepe University Cancer Institute), Altındağ
  - T.C. Saglik Bakanligi - SBU Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Ankara Bilkent City Hospital, Oncology Department, Çankaya
  - Inonu Universitesi - Turgut Ozal Tip Merkezi, Malatya
  - Ondokuz Mayis Universitesi (OMU) - Tip Facultesi, Samsun
  - Medical Park Seyhan Hastanesi, Seyhan
  - T.C. Saglik Bakanligi - Ankara Etlik sehir Hastanesi, Yenimahalle
- United Kingdom (6):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital (AH) - Oncology Centre, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Sarah Cannon Research Institute (SCRI) - London (SCRI-UK), London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital - Sutton, Surrey Quays